CLINICAL TRIAL: NCT00968045
Title: Fibrinogen and Bleeding After Cardiac Surgery
Acronym: Fibro-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Jeppssons, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Fibro 01/07; EudraCT-nr:2007-007157-31
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Complications; Bleeding; Coronary Artery Disease
Keywords: Fibrinogen; Postoperative bleeding; Transfusions; CABG
MeSH Terms: conditions — Hemorrhage; Coronary Artery Disease; Postoperative Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 100 ml infusion of saline is given during 15 minutes after anesthesia induction before start of surgery.
  Interventions: Drug: Fibrinogen
- Study drug (Experimental): Fibrinogen 2g in 100 ml sterile water given during 15 minutes after anestesiainduction before surgery start
  Interventions: Drug: Fibrinogen

INTERVENTIONS:
Drug: Fibrinogen — Fibrinogen 2 gr in 100 ml sterile water. The infusion is given during 15 minutes
  Other Names: Riastap; Haemocomplettan

SUMMARY:
The study hypothesis is that prophylactic fibrinogen infusion reduces postoperative bleeding and transfusion requirements after coronary artery bypass surgery (CABG) in patients with endogenous fibrinogen levels in the lower normal range. 60 patients will be included in a prospective, randomized double-blind placebo-controlled single center study.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age 18 years and above
* Patients eligible for a first-time coronary artery bypass(CABG) surgery with a preoperative fibrinogen plasma concentration under 3,8 g/L
* Signed informed consent to participate in the study

Exclusion Criteria:

* Patients undergoing redo surgery
* Clinical or laboratory signs of bleeding disorder
* Clinical or laboratory signs of significant liver disease, or,other significant disease or condition which in the investigators judgment interfere with hemostasis
* Any medications with agents which may interfere with hemostasis within 14 days prior to study start. Clopidogrel and warfarin are withdrawn at least 24 hours before surgery. Oral aspirin is allowed co-medication.
* Administration of other investigational drugs within eight weeks preceding the preentry examination
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To evaluate safety of prophylactic fibrinogen infusion in patients with fibrinogen levels in the lower normal range undergoing cardiac surgery | 2 years
Blood loss first 12 postoperative hours | 12h

SECONDARY OUTCOMES:
Transfusions | 7 days
Biomarkers of coagulation, fibrinolysis and platelet function | 7 days
Pharmcoeconomic analysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jeppsson, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Cardiothoracic Surgery unit, Sahlgrenska University Hospital, Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Jeppsson A, Walden K, Roman-Emanuel C, Thimour-Bergstrom L, Karlsson M. Preoperative supplementation with fibrinogen concentrate in cardiac surgery: A randomized controlled study. Br J Anaesth. 2016 Feb;116(2):208-14. doi: 10.1093/bja/aev367. Epub 2015 Nov 17. PMID 26577034